CLINICAL TRIAL: NCT06902870
Title: The Effectiveness of a "CARE I DECIDE！" Scenario-Based Online Simulation Training Program in Chest Trauma Care Knowledge and Clinical Reasoning Ability Among Nurses
Brief Title: Effectiveness of Scenario-Based Online Simulation in Chest Trauma in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: tygh backup (Other Government)
Responsible Party: Sponsor-Investigator, tygh backup, Taoyuan General Hospital, Taoyuan General Hospital
Organization: Taoyuan General Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TYGH112053
Record Dates: First submitted 2024-12-17; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Nursing Education
Keywords: Thoracic trauma online simulation clinical reasoning nursing education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group received "Care I Decide!" online simulation-assisted teaching following the classroom-based instruction.
  Classroom-Based Teaching and Online Simulation-Assisted Instruction
  Classroom-Based Instruction:
  Participants were provided with a QR code to access the Moodle platform and download the electronic course materials.
  The classroom instruction covered the following topics:
  Mechanisms of trauma and prehospital assessment. Principles of major trauma activation and evaluation. Types of chest trauma and associated clinical signs. Principles of chest trauma care and recognition of changes in patient conditions.
  "Care I Decide!" Online Simulation-Assisted Teaching:
  A detailed explanation of the operational process for the "Care I Decide!" online simulation-assisted teaching materials was provided.
  The session integrated classroom knowledge with the "Care I Decide!" online simulation. It presented clinical scenarios involving changes in vital signs and symptoms.
  Interventions: Other: Scenario-Based Online Simulation Training Program
- Control Group (Other): The control group received traditional case sharing following the classroom-based instruction.
  Classroom-Based Teaching
  Delivery of Course Materials:
  Participants were provided with a QR code to access the Moodle platform, where they could download the electronic course handouts.
  Classroom Instruction Content:
  The classroom teaching session included the following topics:
  Mechanisms of trauma and prehospital assessment. Principles of major trauma activation and evaluation. Types of chest trauma and associated clinical signs. Principles of chest trauma care and recognition of changes in patient conditions.
  Chest Trauma Case Sharing
  Case Presentation and Reflection:
  Clinical cases involving chest trauma were presented to participants. They were guided to describe the case details, reflect on the management process, and receive constructive feedback.
  Discussion and Problem Solving:
  During the discussion, questions and uncertainties raised by participants were addressed
  Interventions: Other: Classroom-Based Teaching

INTERVENTIONS:
Other: Scenario-Based Online Simulation Training Program — Classroom-Based Teaching and Online Simulation-Assisted Instruction
  Classroom-Based Instruction:
  Participants were provided with a QR code to access the Moodle platform and download the electronic course materials.
  The classroom instruction covered the following topics:
  Mechanisms of trauma and prehospital assessment. Principles of major trauma activation and evaluation. Types of chest trauma and associated clinical signs. Principles of chest trauma care and recognition of changes in patient conditions.
  "Care I Decide!" Online Simulation-Assisted Teaching:
  A detailed explanation of the operational process for the "Care I Decide!" online simulation-assisted teaching materials was provided.
  The session integrated classroom knowledge with the "Care I Decide!" online simulation. It presented clinical scenarios involving changes in vital signs and symptoms of chest trauma patients, guiding participants through clinical decision-making processes.
  Arms: Experimental Group
Other: Classroom-Based Teaching — Classroom-Based Teaching
  Delivery of Course Materials:
  Participants were provided with a QR code to access the Moodle platform, where they could download the electronic course handouts.
  Classroom Instruction Content:
  The classroom teaching session included the following topics:
  Mechanisms of trauma and prehospital assessment. Principles of major trauma activation and evaluation. Types of chest trauma and associated clinical signs. Principles of chest trauma care and recognition of changes in patient conditions.
  Chest Trauma Case Sharing
  Case Presentation and Reflection:
  Clinical cases involving chest trauma were presented to participants. They were guided to describe the case details, reflect on the management process, and receive constructive feedback.
  Discussion and Problem Solving:
  During the discussion, questions and uncertainties raised by participants were addressed to enhance understanding and clarify key concepts.
  Arms: Control Group

SUMMARY:
Methods This randomized controlled trial evaluated teaching strategies for chest trauma education. The course was promoted via posters and conducted over two days, with two sessions per day. Sessions were randomly assigned to the control or experimental group via a lottery system before the course. This process was repeated on day two. A total of 67 participants per group were recruited, ensuring 50% random allocation. Control Group Participants received traditional classroom instruction with case discussions. Pretest: Collected demographic data and assessed baseline knowledge using the Chest Trauma Knowledge Scale (CTKS) and Nursing Clinical Decision-Making Scale (NCDMS). First posttest (1-week follow-up): Measured CTKS, NCDMS, and Learning Engagement Scale (LES). Second posttest (3-month follow-up): Assessed CTKS and Confidence in Nursing Clinical Reasoning Scale (CNCRS). Experimental Group Participants received traditional instruction plus "CARE! I-DECIDE" online simulation. Pretest: Same as the control group. First posttest (1-week follow-up): Measured CTKS, NCDMS, and LES. Second posttest (3-month follow-up): Assessed CTKS and CNCRS. Assessments were completed via Google Forms or paper-based questionnaires. This study compared traditional teaching with blended learning using online simulation, evaluating immediate and delayed outcomes.

DETAILED DESCRIPTION:
Background In Taiwan, accidental injuries remain a major cause of death, with thoracic trauma being a significant contributor to severe cases. Nurses must develop rapid assessment, management, and clinical reasoning skills to improve trauma care. However, trauma training is often limited by spatial and financial constraints, restricting ongoing education. The "Care I Decide!" online simulation-assisted teaching provides a flexible, accessible solution for continuous thoracic trauma training, enhancing nurses' knowledge and clinical reasoning skills.

Purpose This study assessed the effectiveness of "Care I Decide!" in improving nurses' thoracic trauma knowledge and clinical reasoning skills.

Method This randomized controlled trial (RCT) used a two-group, repeated-measures design with 95 ER and surgical nurses from a regional teaching hospital in Northern Taiwan.

* Experimental group (n=49): Received classroom teaching + "Care I Decide!" online simulation.
* Control group (n=46): Received classroom teaching + case sharing.

Participants completed:

* Pre-test (before intervention)
* First post-test (1 week after intervention)
* Second post-test (12 weeks after intervention)

Instruments used:

* Thoracic Trauma Knowledge Scale (TTKS)
* Clinical Reasoning Skills Scale (CRSS)
* Learning Engagement Scale (LES) Results Pre-test scores showed no significant differences between groups.

After the intervention:

* The experimental group had higher thoracic trauma knowledge in both post-tests (p < .01).
* Their clinical reasoning skills improved significantly in the second post-test (p < .05).
* High learning engagement was observed in both groups but was not statistically significant (p > .05).

Conclusion and Recommendations Both approaches improved nurses' knowledge and clinical reasoning skills. The "Care I Decide!" online simulation provided flexible training without time or location constraints. Scenario-based exercises enhanced clinical reasoning and decision-making, offering real-time feedback for concept clarification.

Additionally, interactive videos strengthened knowledge retention and clinical judgment by allowing nurses to apply reasoning in patient scenarios. This method is recommended for continuing education and could be expanded to other trauma scenarios for ongoing clinical training.

ELIGIBILITY:
Inclusion Criteria:

* Professional Setting:

Nurses working in emergency departments or specific surgical specialties, including thoracic surgery, neurosurgery, general surgery, and orthopedics.

Willingness to Participate:

Nurses who voluntarily agree to participate in this study.

Exclusion Criteria:

* Non-Surgical Nurses:

Nurses from non-surgical departments or those not meeting the inclusion criteria within other surgical specialties.

Non-Frontline Care Providers:

Nurses not directly involved in the clinical care of chest trauma patients, such as outpatient nurses or case managers.

Incomplete Participation:

Nurses who do not complete the full course of the study program.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Chest Trauma Knowledge，Clinical Reasoning Scale | 6months
  Primary Outcome Measures: Chest Trauma Care Knowledge Scale：Measures knowledge of chest trauma care.Time Points: Before the intervention, right after the intervention, and 12 weeks later.Clinical Reasoning Scale：Assesses clinical reasoning skills in chest trauma care.Time Points: Before the intervention, right after the intervention, and 12 weeks later.Learning Engagement Scale：Evaluates participants' engagement in the learning process.Time Point: Right after the intervention.Overall Study Time Frame: 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No